CLINICAL TRIAL: NCT02932371
Title: Evaluation of the ECOM™ Monitor for Continuous and Non-invasive Measure of the Cardiac Output in Cardiac Surgery Patients
Acronym: EVALECOM2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2012/11; 2012-A00398-35 (Other: ANSM)
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Cardiac Surgery
Keywords: Cardiac output

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac Surgery (Experimental)
  Interventions: Device: ECOM™.; Device: Trans-esophageal echography

INTERVENTIONS:
Device: ECOM™.
Device: Trans-esophageal echography

SUMMARY:
The objective of the study is to estimate the reliability of the determination of the cardiac output measured by the ECOM™ device. This study will be performed with the latest version of the software which should give better results than those published previously. Two techniques of measure of the cardiac output will be compared: the reference measure by trans-esophageal echography and the bioimpedance used by the ECOM™. monitor.

ELIGIBILITY:
Inclusion Criteria:

* Patients over18 years
* Needed cardiac surgery,
* Needed a monitoring by transesophageal ultrasound ,
* Benefiting from a social security scheme
* Having given their written consent.

Exclusion Criteria:

* Pregnant or breast-feeding women,
* Allergy to polyvinylchloride (PVC),
* The patients for whom a difficulty of ventilation with a mask or intubation is envisaged,
* Contraindication to transesophageal ultrasound, a steady cardiac arrhythmia, a flight or an aortic shrinkage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Cardiac output | 4 hours

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Chirurgical Marie-Lannelongue, Le Plessis-Robinson
  - Institut Mutualiste Montsouris, Paris

IPD SHARING:
Plan to Share IPD: No